CLINICAL TRIAL: NCT06433479
Title: Efficacy of DApagliflozin on REcurrence After Catheter Ablation for Atrial Fibrillation
Acronym: DARE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-4-20610
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation; Atrial fibrillation; Recurrence; Dapagliflozin; AF Burden
MeSH Terms: conditions — Atrial Fibrillation; Recurrence | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg per day for 3 months after initial catheter ablation
  Interventions: Drug: Dapagliflozin 10 mg per day for 3 months after initial catheter ablation
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Dapagliflozin 10 mg per day for 3 months after initial catheter ablation — Dapagliflozin 10 mg per day for 3 months after initial catheter ablation
  Arms: Dapagliflozin

SUMMARY:
This is a single-center, parallel-group, randomized, open-label trial evaluating the effect of 3-month treatment with dapagliflozin 10mg once daily on the recurrence of atrial fibrillation after catheter ablation for atrial fibrillation in patients without diabetes, heart failure, or chronic kidney disease.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common arrhythmias. Catheter ablation of atrial fibrillation, as the main means of rhythm control, can effectively maintain sinus rhythm, reduce the recurrence of AF burden, and improve the patient's quality of life and prognosis. However, AF recurrence still occurs in 30-50% of patients after atrial fibrillation catheter ablation, and there is currently no effective strategy to reduce the recurrence rate after atrial fibrillation ablation.

Sodium-glucose cotransporter 2 inhibitors (SGLT2i) are a new class of diabetic drugs and large clinical trials have established their multiple cardiovascular benefits. Several studies demonstrated that SGLT2i might reduce AF/atrial flutter events among patients with diabetes. Our cohort study and meta-analysis demonstrated a lower risk of AF recurrence with the use of SGLT2i among patients with diabetes after AF ablation. However, the beneficial effects of SGLT2i in patients after AF catheter ablation without current indications for SGLT2i were uncertain.

In this study, we aim to evaluate the effect of dapagliflozin on AF burden. Patients with persistent AF undergoing initial catheter ablation without diabetes at high cardiovascular risk, heart failure, or chronic kidney disease will be enrolled. Patients will be randomly assigned to either the dapagliflozin group (10mg/d) for 3 months or the control group stratified according to body mass index (<24, ≥24kg/m2) or left atrial diameter (<45，≥45mm).

The primary outcome is atrial fibrillation burden calculated as the percentage of of all atrial arrhythmia episodes detected by 7-day single-lead ECG patches at 3 months after ablation. Quality of life and echocardiography changes of left atrial structure will also be evaluated at 3 months. Our central hypothesis is that SGLT2i will reduce the AF burden after catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-80 years
2. diagnosed with persistent atrial fibrillation based on ECG or Holter
3. planned initial catheter ablation for atrial fibrillation
4. have the capacity to understand and sign an informed consent form.

Exclusion Criteria:

1. diagnosed with persistent atrial fibrillation longer than 5 years or left atrial anterior-posterior diameter ≥ 50mm
2. diagnosed with atrial fibrillation secondary to reversible causes (such as hyperthyroidism, acute infection, etc.)
3. severe structural heart disease (hypertrophic cardiomyopathy, rheumatic heart disease, dilated cardiomyopathy, etc.)
4. currently take sodium-glucose co-transporter 2 inhibitors
5. have the following Class I indications for sodium-glucose co-transporter 2 inhibitors: i. type 2 diabetes ii. history of heart failure (HF), including HF with reduced ejection fraction, mildly reduced ejection fraction, and preserved ejection fraction iii. chronic kidney disease with eGFR=20-60 ml/min/1.73m2
6. have the following contraindication of sodium-glucose co-transporter 2 inhibitors: i. previous allergic reactions to dapagliflozin ii. end-stage renal failure or dialysis
7. type 1 diabetes, or previous diabetic ketoacidosis
8. severe hypoglycemia or genitourinary infection in the past 12 months
9. hypovolemia or hypotension
10. planned surgery or other interventional procedure within 3 months
11. other arrhythmias mandating anti-arrhythmic drug therapy
12. have intracardiac thrombus
13. active infection
14. unable to give informed consent
15. women of childbearing potential
16. currently enrolled in another clinical study
17. other condition unsuitable to participate in this study judged by investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation burden at 3 months after ablation | 3 months
  Atrial fibrillation burden is defined as the percent of time spent in atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) episodes detected by 7-day single-lead ECG patches at 3 months after ablation.

SECONDARY OUTCOMES:
Atrial fibrillation recurrence during 3 months after ablation | 3 months
  Atrial fibrillation recurrence is defined as the first recurrence of any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) lasting 30 seconds or longer detected by ECG during 3 months after ablation.
Changes of quality of life at 3 months | 3 months
  Changes of quality of life from baseline to 3 months after ablation evaluated by the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire.
Echocardiography changes of left atrial structure at 3 months | 3 months
  Changes in the echocardiography parameter of anteroposterior atrial diameter from baseline to 3 months after ablation.
Atrial fibrillation recurrence during 1 year after ablation | 1 year
  Atrial fibrillation recurrence is defined as the first recurrence of any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) lasting 30 seconds or longer detected by ECG during 1 year after ablation.
Cardiovascular outcomes during 1-year follow-up | 1 year
  The composite endpoint of cardiovascular death or cardiovascular hospitalization during 1-year follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang C, Zhao Z, Yang Z, Wang Y, Xu Y, Xu H, Guo H, Wang C, He L, Xia S, Kong X, Dai W, Zhang J, Zuo S, Liu X, Guo X, Liu N, Li S, Zhou N, Jiang C, Tang R, Sang C, Zei PC, Long D, Du X, Dong J, Macle L, Ma C. Dapagliflozin to Reduce Early Recurrence After Catheter Ablation for Atrial Fibrillation: The DARE-AF Randomized Clinical Trial. Circulation. 2026 Feb 3;153(5):297-306. doi: 10.1161/CIRCULATIONAHA.125.077447. Epub 2025 Nov 9. PMID 41206792